CLINICAL TRIAL: NCT06105268
Title: The Effect of a Flipped Learning Approach on Midwifery Students Learning Shoulder Dystocia Management: A Randomized Controlled Trial.
Brief Title: Management of Shoulder Dystocia in Flipped Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Reyhan Aydin Doğan, Assistant professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022/1141
Record Dates: First submitted 2023-10-16; First posted 2023-10-27 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-01

CONDITIONS: Shoulder Dystocia - Delivered
Keywords: Shoulder Dystocia; flipped learning; midwifery student
MeSH Terms: conditions — Shoulder Dystocia

STUDY DESIGN:
Intervention Model Description: The sample of the study will consist of two groups: experimental and control. The number of students in each group is the difference between the experimental and control groups in order to determine the effectiveness of shoulder dystocia management given using the flipped learning technique; With 95% confidence (1-α), 95% test power (1-β), d = 1.3000000 effect size and two-sided t test, the number of samples to be taken in each group will be 17 and the study should be conducted with a total of 34 students (16). . Since there is no case of data loss and there is no sample study where the flipped learning technique and shoulder dystocia are used together, a total of 68 students will be studied, 34 students in each group.
Who Masked: Investigator
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- flipped learning group (Experimental): In addition to the traditional theory training to be given within the scope of the study, two hours of video-supported shoulder dystocia training will be given using the university's corporate Microsoft teams program, one day before the simulation application. The videos used in the training consist of previously shot training videos. There is no copyright or legal problem in using the videos.
  Interventions: Other: flipped learning training group
- routine training group- control group (No Intervention): The control group will be given shoulder dystocia theory training before the simulation training within the routine course protocol within the scope of the routine risky birth and postpartum period course.

INTERVENTIONS:
Other: flipped learning training group — flipped learning training group. Applying a flipped learning model in addition to routine training in a fully equipped simulation
  Arms: flipped learning group

SUMMARY:
Flipped learning is an innovative learning method in midwifery education. Studies that apply this learning method together with shoulder dystocia training have not been found in the current literature. For this reason, the study was designed as a randomized controlled study to examine the effectiveness of the flipped learning technique in shoulder dystocia management using high-valid simulation in midwifery undergraduate education.

DETAILED DESCRIPTION:
Flipped learning is an innovative learning method in midwifery education. Studies that apply this learning method together with shoulder dystocia training have not been found in the current literature. For this reason, the study was designed as a randomized controlled study to examine the effectiveness of the flipped learning technique in shoulder dystocia management using high-valid simulation in midwifery undergraduate education.

Hypotheses of the research;

First Hypothesis H1: The use of flipped learning model in midwifery education has an effect on midwifery students' shoulder dystocia knowledge levels.

Second Hypothesis H1: The use of flipped learning model in midwifery education has an effect on midwifery students' levels of Student Satisfaction and Self-Confidence in Learning.

Third Hypothesis H1: The use of flipped learning model in midwifery education has an effect on midwifery students' Pagana Clinical Stress levels.

ELIGIBILITY:
Inclusion Criteria:

* - Agreeing to participate in the study,
* Being a 4th year student at the Department of Midwifery,

Exclusion Criteria:

* - Refusing to participate in the study,
* Being a 1st, 2nd and 3rd year student in the midwifery department

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
H1 | 12 months
  Using the flipped learning model in midwifery education increases the knowledge level score of midwifery students on shoulder dystocia.
H1 | 12 months
  Using the flipped learning model in midwifery education reduces the PANAGA clinical stress level score of midwifery students.
H1 | 12 months
  Using the flipped learning model in midwifery education increases midwifery students' oStudent Satisfaction and Self-Confidence in Learning Scale scores.

OTHER OUTCOMES:
Measurement and evaluation materials to be used in the study | Scales will be administered immediately after the educational intervention.
  In the study, a personal data form containing students' personal information,
Measurement and evaluation materials to be used in the study | Scales will be administered immediately after the educational intervention.
  Shoulder Dystocia and Management Information Form
Measurement and evaluation materials to be used in the study | Scales will be administered immediately after the educational intervention.
  Shoulder Dystocia Management Individual Evaluation Form will be used to determine the effectiveness of the training.
Measurement and evaluation materials to be used in the study | Scales will be administered immediately after the educational intervention.
  The Student Satisfaction and Self-Confidence Scale in Learning will be used to determine students' simulation competencies and satisfaction,
Measurement and evaluation materials to be used in the study | Scales will be administered immediately after the educational intervention.
  The Pagana Clinical Stress Survey will be used to determine the stress caused by application techniques on students.

CONTACTS AND LOCATIONS:
Locations (1):
- Reyhan Aydin Doğan, Karabük, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It will be shared when the work is completed.

REFERENCES:
- [Background] Saritas E, Baykara ZG. The effect of flipped learning approach on nursing students' learning of patient safety: A randomized controlled trial. Nurse Educ Pract. 2023 Oct;72:103742. doi: 10.1016/j.nepr.2023.103742. Epub 2023 Aug 10. PMID 37611355
- [Background] Golaki SP, Kamali F, Bagherzadeh R, Hajinejad F, Vahedparast H. The effect of Flipped Classroom through Near Peer Education (FC through NPE) on patient safety knowledge retention in nursing and midwifery students: a solomon four-group design. BMC Med Educ. 2022 Feb 19;22(1):112. doi: 10.1186/s12909-022-03144-w. PMID 35183160
- See also: Flipped Classroom Learning Experiences of Graduate Nursing Students in Advanced Pathophysiology and Pharmacology in Midwifery Course — https://medicopublication.com/index.php/ijone/article/view/3696